CLINICAL TRIAL: NCT00084435
Title: Adjuvant Chemo-RT With Cisplatin (NSC-119875) and Docetaxel (NSC-628503) After Complete Resection of Locally Advanced (Stage III and IV) Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: S0217, Adjuvant Cisplatin and Docetaxel After Complete Resection Stage III or IV Head and Neck Cancer
Acronym: S0217
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and suspension of head and neck committee
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365311; S0217 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III salivary gland cancer; stage IV salivary gland cancer; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; salivary gland squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemoRT after surgery (Experimental): chemoRT with cisplatin and docetaxel after surgery
  Interventions: Drug: cisplatin; Drug: docetaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin — 75 mg/m2 IV, Day 1, q 21 days for 3 cycles
  Other Names: platinol
Drug: docetaxel — 15 mg/m2 IV, Day 1, 1 7 days for 6 doses
  Other Names: taxotere
Radiation: radiation therapy — 200 cGy/day, Days 1-5, q week for 6 weeks
  Other Names: RT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Cisplatin and docetaxel may make the tumor cells more sensitive to radiation therapy. Giving chemoradiotherapy after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well adjuvant chemoradiotherapy using cisplatin and docetaxel works in treating patients with completely resected stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the disease-free survival and overall survival of patients with high-risk stage III or IV squamous cell carcinoma of the head and neck treated with adjuvant chemoradiotherapy comprising docetaxel and cisplatin.
* Determine the toxicity of this regimen in these patients.
* Categorize the site(s) of disease relapse in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on days 1, 8, 15, 22, 29, and 36 and cisplatin IV over 1.5 hours on days 1, 22, and 43. Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-45. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 3 years from registration.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study within 17.5-23.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of squamous cell carcinoma of the head and neck

  * Selected stage III or IV (no distant metastasis) disease

    * The following TNM stages are excluded:

      * T3, N0, M0
      * T4a, N0, M0
      * T4b, N3, M0
      * Any T, any N, M1
* Complete total resection within the past 56 days AND has one or more of the following risk factors:

  * Multiple pathologically confirmed lymph node metastases
  * One or more lymph nodes with extracapsular extension of tumor
  * Microscopically positive margin(s) of resection, including mucosal margins and/or soft tissue or deep margins of resection
* No primary nasopharyngeal carcinoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Other

* No pre-existing peripheral neuropathy
* No known history of severe hypersensitiviy reaction to products containing Polysorbate 80
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for the malignancy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for the malignancy

Surgery

* See Disease Characteristics

Other

* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Disease progression
Disease-free survival
Symptomatic deterioration
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Prakash C. Neupane, MD, Principal Investigator — St. Mary's Cancer Specialists at St. Mary's Health Center; Harold E. Kim, MD, Study Chair — Barbara Ann Karmanos Cancer Institute; Stephen K. Williamson, MD, Study Chair — University of Kansas; George H. Yoo, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (29):
- United States (29):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina